CLINICAL TRIAL: NCT05371262
Title: Evaluation of Long-term Benefit-risk Profile of Levothyroxine Treatment in Children With Congenital Hypothyroidism: Influence of Initial Levothyroxine Dose on Neurodevelopmental, Growth, Cardiovascular and Skeletal Outcomes
Brief Title: Influence of Initial Levothyroxine Dose on Neurodevelopmental and Growth Outcomes in Congenital Hypothyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof.ssa Mariacarolina Salerno, Associate Professor of Pediatrics, Head of Pediatric Endocrinology Unit, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FARM8A8FHP
Record Dates: First submitted 2022-05-04; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Congenital Hypothyroidism
Keywords: Neonatal screening; Levothyroxine treatment; Neurocognitive; Growth
MeSH Terms: conditions — Congenital Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: Children were randomly assigned to receive an initial L-T4 dose of 10-12.5 μg/kg/day (Group A) or 12.6-15 μg/kg/day (Group B). Randomization was designed according to a block scheme (8 blocks of 6 patients and 6 blocks of 4 patients which were randomly alternated) which guaranteed the frequency balance in the two groups during the enrolment without altering the causality of the assignment. Random allocation sequence was generated using the function sample in R statistical platform.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10-12.5 μg/kg/day of L-T4 (Active Comparator): Children with congenital hypothyroidism who received an initial L-T4 dose of 10-12.5 μg/kg/day.
  Interventions: Drug: Levothyroxin
- 12.6-15 μg/kg/day of L-T4 (Active Comparator): Children with congenital hypothyroidism who received an initial L-T4 dose of 12.6-15 μg/kg/day.
  Interventions: Drug: Levothyroxin

INTERVENTIONS:
Drug: Levothyroxin — Congenital hypothyroidism children received two different doses of levothyroxin within the recommended range to evaluate any differences in long-term outcomes.
  Other Names: L-T4

SUMMARY:
The primary objective of this study is to evaluate the risk-benefit profile of long-term treatment of two different initials treatment schemes with L-T4 on the neurodevelopmental and auxological outcomes in children with congenital hypothyroidism, diagnosed by neonatal screening in order to find the best dose of initial thyroid hormone replacement to assure the best long-term developmental outcome without any adverse effects on auxological, cardiovascular and skeletal outcomes. The secondary objective of the study is to evaluate the role of other factors that, in addition to the initial L-T4 therapy,can influence long-term neurodevelopmental and auxological outcomes as well as the cardiovascular system and bone metabolism outcomes.

DETAILED DESCRIPTION:
Seventy-two neonates detected by the neonatal screening program for congenital hypothyroidism were randomly assigned to receive one of the two initial L-T4 replacement dose: Group A received an initial replacement dose of 10-12.5 mcg/kg/die and Group B received an initial replacement dose of 12.6-15 mcg/kg/die. The adequacy of treatment were monitored closely by clinical evaluation and regular measurement of FT4 and TSH. Cognitive development were evaluated through the Griffiths Mental Development Scales at the the age of 2 yeas. Cognitive and behavioural assessment at the age of 4 years were performed using the Wechsler Preschool and Primary scale of Intelligence. Growth were evaluate at the enrolment and at each visit. Skeletal maturation were evaluated at diagnosis and at the age of 1 and 4 years. At the age of 4 years a quantitative ultrasound measurements and cardiovascular evaluation were performed.

ELIGIBILITY:
Inclusion Criteria:

* Congenital Hypothyroidism diagnosed by neonatal screening program
* Age less than 30 days at diagnosis
* TSH value at confirmatory diagnosis above 30 mU/l
* Caucasian ethnicity

Exclusion Criteria:

* Prematurity
* Major congenital malformations
* Neonatal diseases
* Chromosomopathies
* Known maternal thyroid diseases

Ages: 3 Days to 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental outcomes | At four years of age
  Cognitive and behavioral assessment was performed using Wechsler Preschool and Primary scale of Intelligence (WIPPSI-III). The WIPPSI-III evaluates the intelligence of children between 2.6 and 7.3 years and provides a Total Intelligence Quotient, a Verbal Intelligence Quotient, a Performance Intelligence Quotient and a Processing Speed Quotient. Quotients > 85 are considered normal.
Linear Growth | 7-10 days after the start of treatment and at 1.5, 3, 6, 9, 12, 18, 24, 30, 36, 42 and 48 months of life.
  Linear growth was evaluated periodically during the study through the measurement of length up to 3 years and height subsequently. Length and height were measured in centimeters and are expressed as standard deviation score.

CONTACTS AND LOCATIONS:
Overall Officials: Mariacarolina Salerno, Professor, Principal Investigator — Federico II University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leger J, Olivieri A, Donaldson M, Torresani T, Krude H, van Vliet G, Polak M, Butler G; ESPE-PES-SLEP-JSPE-APEG-APPES-ISPAE; Congenital Hypothyroidism Consensus Conference Group. European Society for Paediatric Endocrinology consensus guidelines on screening, diagnosis, and management of congenital hypothyroidism. J Clin Endocrinol Metab. 2014 Feb;99(2):363-84. doi: 10.1210/jc.2013-1891. Epub 2014 Jan 21. PMID 24446653
- [Background] American Academy of Pediatrics; Rose SR; Section on Endocrinology and Committee on Genetics, American Thyroid Association; Brown RS; Public Health Committee, Lawson Wilkins Pediatric Endocrine Society; Foley T, Kaplowitz PB, Kaye CI, Sundararajan S, Varma SK. Update of newborn screening and therapy for congenital hypothyroidism. Pediatrics. 2006 Jun;117(6):2290-303. doi: 10.1542/peds.2006-0915. PMID 16740880
- [Background] Ng SM, Anand D, Weindling AM. High versus low dose of initial thyroid hormone replacement for congenital hypothyroidism. Cochrane Database Syst Rev. 2009 Jan 21;2009(1):CD006972. doi: 10.1002/14651858.CD006972.pub2. PMID 19160309
- [Derived] Esposito A, Vigone MC, Polizzi M, Wasniewska MG, Cassio A, Mussa A, Gastaldi R, Di Mase R, Vincenzi G, Pozzi C, Peroni E, Bravaccio C, Capalbo D, Bruzzese D, Salerno M. Effect of initial levothyroxine dose on neurodevelopmental and growth outcomes in children with congenital hypothyroidism. Front Endocrinol (Lausanne). 2022 Sep 5;13:923448. doi: 10.3389/fendo.2022.923448. eCollection 2022. PMID 36133316